CLINICAL TRIAL: NCT00096616
Title: A Single Dose, Randomized, Double-blind Crossover Comparison of Combivent CFC MDI and Albuterol HFA MDI in Patients With Moderate to Severe Persistent Asthma and Persistent Symptoms Despite Treatment With Inhaled Corticosteroids
Brief Title: Combivent® CFC Metered Dose Inhaler (MDI) in Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.50
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Combivent® CFC MDI
Drug: Albuterol HFA MDI

SUMMARY:
The purpose of this study is to demonstrate the superior bronchodilator efficacy of inhaled Combivent® CFC MDI vs. Albuterol HFA MDI in moderate to severe asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than or equal to 18 years of age,
* non-smokers,
* diagnosed with asthma, with an FEV1 less than or equal to 70 percent of predicted normal,
* stable use of Beta agonist
* daily use of inhaled steroids for one year

Exclusion Criteria:

* Patients with other significant diseases other than asthma, requiring oxygen,
* intubated within 5 years,
* asthma exacerbation within 6 weeks of trial,
* use of unstable doses (greater than 10 mg/day of prednisone or equivalent) of steroids,
* participating in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-11; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
FEV1 area under the curve (AUC) 0 to 6 hours Peak FEV1

SECONDARY OUTCOMES:
FEV1 at each timepoint Peak FVC FVC at each timepoint FVC AUC 0-6 Adverse events Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (27):
- United States (27):
  - 620 South 20th Street, NHB 104, Birmingham, Alabama
  - Cooper Green Hospital, Birmingham, Alabama
  - Southern California Clinical Trials, Lakewood, California
  - Boehringer Ingelheim Investigational Site, Palmdale, California
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Panama City, Florida
  - Boehringer Ingelheim Investigational Site, Coeur d'Arlene, Idaho
  - Boehringer Ingelheim Investigational Site, River Forest, Illinois
  - Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - LSU MC-Sheveport, Shreveport, Louisiana
  - Boehringer Ingelheim Investigational Site, Auburn, Maine
  - Johns Hopkins Asthma & Allergy, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boehringer Ingelheim Investigational Site, Berlin, New Jersey
  - Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU School of Medicine, New York, New York
  - Division of Pulmonary & Critical Care Medicine, Durham, North Carolina
  - Wake Forest University, Center for Human Genomics, Winston-Salem, North Carolina
  - Penn State University, Hershey Medical Center, Hershey, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Ben Taul General Hospital, Houston, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - University of Wisconsin Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Gelb AF, Karpel J, Wise RA, Cassino C, Johnson P, Conoscenti CS. Bronchodilator efficacy of the fixed combination of ipratropium and albuterol compared to albuterol alone in moderate-to-severe persistent asthma. Pulm Pharmacol Ther. 2008 Aug;21(4):630-6. doi: 10.1016/j.pupt.2008.02.005. Epub 2008 Mar 5. PMID 18403223